CLINICAL TRIAL: NCT01276626
Title: Pilot Study of Probiotic Bifidobacterium Longum (B. Longum) on Mood and Bowel Symptoms in Patients With Irritable Bowel Syndrome (IBS).
Brief Title: Study of Bacteria on Mood and Bowel Symptoms in Patients With Irritable Bowel Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Nestle 09.25.NRC
Record Dates: First submitted 2010-12-27; First posted 2011-01-13 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Irritable Bowel Syndrome; IBS
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bifidobacterium longum (Experimental)
  Interventions: Dietary Supplement: Bifidobacterium longum
- Maltodextrin (Placebo Comparator)
  Interventions: Other: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Bifidobacterium longum — Powder containing Bifidobacterium longum in maltodextrin.
  Arms: Bifidobacterium longum
Other: Maltodextrin — Powder containing only maltodextrin
  Arms: Maltodextrin

SUMMARY:
The purpose of this study is to determine whether probiotic bacterium Bifidobacterium longum (B. longum) can improve mood and bowel symptoms in patients with Irritable bowel syndrome (IBS). The patients will be treated with probiotic or placebo for 6 weeks. Their mood, memory, general well-being and bowel symptoms will be assessed before, at the end of the treatment and 4 weeks later. Brain activation pattern, changes in gut bacteria, metabolic profile and inflammatory markers will be also measured.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Irritable Bowel Syndrome based on Rome III Criteria
* Symptoms of mild to moderate anxiety and depression

Exclusion Criteria:

* Concurrent systemic disease and/or laboratory abnormalities considered by Investigators to be risky or that could interfere with data collection.
* Concurrent organic Gastrointestinal (GI) pathology other than benign polyps, diverticulosis, hemorrhoids, lipomas and melanosis coli.
* Psychiatric diagnosis other than anxiety or depression.
* Patients treated with therapeutic/standard doses of antidepressants and/or anxiolytics
* History of active cancer in the last 5 years, other than skin basal cells cancer
* Pregnant or breastfeeding women
* Treatment with antibiotics during the three months prior the study.
* Known or suspected allergies to the study products (eg maltodextrin).
* Patients who have heart pacemakers, metal implants, metal chips or clips in or around the eyeballs, artificial heart valves, metallic ear implants, bullet fragments or fixed brackets.
* High fiber diet (>35 g/day for males, > 25 g/day for females), consumption of high inulin containing foods (>5 g/day).
* Consumption of any type of yoghurts or probiotic-containing products in the 4 weeks prior to the beginning of the study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression (HAD) scale. | 6 weeks post-treatment initiation
  Change in anxiety and depression, assessed using Hospital Anxiety and Depression (HAD) scale, after six weeks of treatment.

SECONDARY OUTCOMES:
Improvement in IBS symptoms. | 6 and 10 weeks post-treatment
Improvement in objective biomarkers. | 6 weeks post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Peter McLean, PhD, Study Director — Société des Produits Nestlé (SPN); Premysl Bercik, MD, Principal Investigator — McMaster University
Locations (1):
- McMaster University Medical Center, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Pinto-Sanchez MI, Hall GB, Ghajar K, Nardelli A, Bolino C, Lau JT, Martin FP, Cominetti O, Welsh C, Rieder A, Traynor J, Gregory C, De Palma G, Pigrau M, Ford AC, Macri J, Berger B, Bergonzelli G, Surette MG, Collins SM, Moayyedi P, Bercik P. Probiotic Bifidobacterium longum NCC3001 Reduces Depression Scores and Alters Brain Activity: A Pilot Study in Patients With Irritable Bowel Syndrome. Gastroenterology. 2017 Aug;153(2):448-459.e8. doi: 10.1053/j.gastro.2017.05.003. Epub 2017 May 5. PMID 28483500